CLINICAL TRIAL: NCT00911742
Title: Comparative Bioavailability Between Two Tramadol Formulations: Study of the Better Controlled Release of a New 200 mg OAD Formulation Versus Zytram® 200 mg
Brief Title: Comparative Bioavailability Between Two Tramadol Formulations: Study of the Better Controlled Release of a New 200 mg Once A Day (OAD) Formulation Versus Zytram® 200 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Vice-President Regulatory Affairs, Labopharm Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MDT1-012
Record Dates: First submitted 2009-04-08; First posted 2009-06-02 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Tramadol

ARMS (2):
- 1 Tramadol Contramid Once A Day (Experimental)
  Interventions: Drug: Tramadol Contramid OAD
- 2 Zytram (R) (Active Comparator)
  Interventions: Drug: Zytram

INTERVENTIONS:
Drug: Tramadol Contramid OAD — 1 Tramadol Contramid OAD 200 mg tablet as a single dose
  Arms: 1 Tramadol Contramid Once A Day
Drug: Zytram — 1 Zytram 200 mg tablet as a single dose
  Arms: 2 Zytram (R)

SUMMARY:
The main purpose of this study is to compare the pharmacokinetic profile to establish the better controlled liberation of the test product (Tramadol HCL OAD tablets of 200 mg, Labopharm) and its bioavailability in relation with the commercialised reference (Zytram® tablets of 200 mg, Zambon), single dose administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of either gender
* Age between 18 and 45 years
* Body mass index between 19 and 27kg/m2
* Normal medical history
* Normal or no clinically significant physical examination findings
* Normal or no clinically significant findings in analytical tests
* Negative hepatitis B, hepatitis C or HIV serology
* Negative drugs of abuse in urine
* Negative pregnancy test in females
* The subject understands and accepts the study procedures and grants in writing his/her informed consent

Exclusion Criteria:

* Did not fulfill the inclusion criteria
* Organic disorders or underwent major surgery, within 90 days before study screening
* Psychiatric history
* Alcohol drink intake greater than 30gr/day
* Cigarette smoking greater than 10 cigarettes/day
* Excessive consumption of food or beverages containing xanthines (more than five units of coffee, tea or cola per day)
* Medical treatment within 30 days before screening, and/or any medication 7 days before starting the study
* Participation in other clinical study or donate blood within 90 days before starting this study
* Antecedents of gastric, hepatic, renal and other kind of disorder that could affect ADME (absorption, distribution, metabolism or excretion of the study drug)
* Hepatitis B, hepatitis C or HIV positive serology
* Pregnant or breastfeeding
* Clinically relevant hypersensitivities (in particular to drugs)
* Woman taking oral contraceptive drugs
* Incapable of communicating and cooperating with investigators

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2004-02; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

REFERENCES:
- [Result] Hernandez-Lopez C, Martinez-Farnos L, Karhu D, Perez-Campos T, Rovira S, Encina G. Comparative bioavailability between two Tramadol once-daily oral formulations. Methods Find Exp Clin Pharmacol. 2006 Jul-Aug;28(6):373-8. doi: 10.1358/mf.2006.28.6.1007674. PMID 16894407

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol Contramid Once A Day: Single oral administration of 1x200mg Tramadol OAD tablet according to randomization schedule. There were 2 treatment sequences, each separated by at least one week wash-out period.
  OAD: Once-A-Day
- Zytram (R): Single oral administration of 1x200mg Zytram tablet according to randomization schedule. There were 2 treatment sequences, each separated by at least one week wash-out period.
  OAD: Once-A-Day
Period: Treatment Phase I
Arm/Group | Tramadol Contramid Once A Day | Zytram (R)
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Treatment Phase II
Arm/Group | Tramadol Contramid Once A Day | Zytram (R)
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol Contramid Once A Day | Zytram (R) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 13 | 13 | 26.0
  >=65 years | 0 | 0 | 0.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13.0
  Male | 8 | 5 | 13.0

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-t)
Description: Area under the plasma concentration versus time curve to the last measured concentration.
  h=hour
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Tramadol Contramid Once A Day | Zytram (R)
Number analyzed (Participants) | 26 | 26
ng.h/mL | 5886 (1843) | 4761 (1623)

2. Primary Outcome: AUC (0-∞)
Description: The area under the plasma concentration curve was estimated by extrapolating to infinity AUC0-t. The extrapolation to infinity was done by regression with the last log-transformed data to estimate the terminal area by means of the line that maximized R'2 (coefficient of determination). The units are ng.h/mL.
  h=hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Tramadol Contramid Once A Day | Zytram (R)
Number analyzed (Participants) | 26 | 26
ng.h/mL | 6112 (2078) | 5638 (2274)

3. Primary Outcome: Cmax
Description: Maximum plasma concentration
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tramadol Contramid Once A Day | Zytram (R)
Number analyzed (Participants) | 26 | 26
ng/mL | 270 (96) | 219 (50)

4. Secondary Outcome: t1/2
Description: Apparent terminal elimination half-life
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tramadol Contramid Once A Day | Zytram (R)
Number analyzed (Participants) | 26 | 26
hours | 7.41 (2.15) | 14.92 (7.11)

5. Secondary Outcome: Tmax
Description: Time to maximum plasma concentration
Time Frame: 48 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Tramadol Contramid Once A Day | Zytram (R)
Number analyzed (Participants) | 26 | 26
hours | 9.0 [2 to 16] | 4.5 [2 to 12]

ADVERSE EVENTS:
Arm/Group | Tramadol Contramid Once A Day | Zytram (R)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 8/26 | 9/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Contramid Once A Day (N=26) | Zytram (R) (N=26)
Headache (General disorders) | 1 | 2
Somnolence (Psychiatric disorders) | 2 | 2
Dizziness (Nervous system disorders) | 6 | 4
nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must agree to maintain the confidentiality of the study at all times, and he cannot reveal any information coming from the protocol, the study results or any documentation related to the study, without permission of the sponsor. Any publication of the results, in whole or in part will require the permission of the sponsor.